CLINICAL TRIAL: NCT07112638
Title: Effects of an Immersive Technology-based Intergenerational Intervention to Improve Movement Patterns in Older Adults: Co-creation and a Randomised Controlled Trial (engAGE) Study Protocol.
Brief Title: The engAGE Project: Immersive Intergenerational Intervention to Improve Movement in Older Adults
Acronym: engAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PID2022-140660NB-C21; PID2022-140660NB-C21 (Other Grant/Funding Number: Ministerio de ciencia, innovación y universidades - España)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Frailty at Older Adults
Keywords: co-creation; intergenerational; physical activity; sedentary behavior; older adults
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Immersive virtual reality + exercise (Experimental): Intervention: Immersive virtual reality + phisical exercises
  Interventions: Other: immersive technology-based intergenerational intervention to improve movement patterns in older adults
- Control (No Intervention): workshops including story telling, origami and yoga

INTERVENTIONS:
Other: immersive technology-based intergenerational intervention to improve movement patterns in older adults — Intervention group The intervention consists of 60-minute supervised sessions conducted once per week for 12 weeks. Each session begins with a 10-minute warm-up, followed by 15 minutes of strength training. Four structured session types (A, B, C, and D) were designed and are being rotated throughout the 12-week period. These sessions incorporate upper and lower body exercises performed using body weight and/or resistance bands, adapted to each participant's physical function.
  Arms: Intervention: Immersive virtual reality + exercise

SUMMARY:
The engAGE project is an innovative, non-oriented research initiative that seeks to advance public health knowledge to promote quality of life and functional independence in older adults. It combines expertise in public health, education, pedagogy, psychology, and technology with a novel approach.

The project is divided in two phases:

Phase 1:

Involves the co-creation of an intergenerational intervention designed to improve movement patterns of community-dwelling older adults (65+), recruited from community and day care centres. Using participatory action research, interventions will be co-designed with older adults, family members (including children and grandchildren), students, health and education professionals, technology experts, and researchers. The reserachers aim is to reduce sedentary behaviour (SB), increase physical activity (PA), and explore the added value of immersive technology to enhance uptake, adherence, and sustainability.

Phase 2:

Evaluate the effects of the tailored, co-created intervention through a randomised controlled clinical trial. Movement patterns will be assessed via accelerometry and observational measures (time in SB, active vs. passive SB, standing, walking, steps, and transitions) at baseline, post-intervention, 6 months, and 12 months. In addition to movement outcomes, secondary measures will include functional capacity, independence, loneliness, social isolation, physical function, body composition, quality of life, depression, anxiety, and cost-utility.

DETAILED DESCRIPTION:
The present project is innovative, and it is presented as a non-oriented research project that aims to advance the current knowledge of promoting public health research for a better quality of life and functional independence of the older adult population, including community-dwelling older adults. The current proposal brings together knowledge in public health, education, pedagogy, psychology, and technology with a novel approach.

The EngAGE project approaches to co-create an intergenerational intervention aimed at improving PA and reducing SB in community-dwelling older adults, followed by an evaluation of its effects on PA and SB, with a special focus on whether these effects are maintained in the mid and long term.

The project is divided in two phases:

Phase 1:

Co-create an intergenerational intervention based on technology solutions to improve movement patterns [reduce sedentary behaviour (SB) and increase physical activity (PA) levels] of community-dwelling older adults (recruited from day care and community centres) (65 years and older). Tailored to each setting, interventions will be designed together with end-users, family members (including children and grandchildren), primary and secondary school students, health professionals, health management professionals (e.g., hospital directors), technology experts, primary and secondary education professionals (teachers), researchers, and sport sciences specialists to reduce SB and increase PA levels of older adults through participatory action research methodology, specifically co-creation. The investigators also aim to explore the added value of immersive technology to increase and enhance uptake, adherence, and sustainability of an intervention to improve movement patterns in the older adult population.

Phase 2:

To evaluate the effects of the intervention programs, tailored to each setting, co-created in Phase 1 on the movement patterns (time in SB, time in mentally active and passive SB, standing time, walking time, number of steps, number and time of transitions) of older adults (65 years and older) in the short (end of intervention), medium and long term (with 6 and 12 months post-intervention follow-up, respectively), by means of a randomised controlled clinical trial. As secondary objectives, the investigators intend to evaluate the effects of the intervention programs on functionality/dependence, loneliness and social isolation, physical function, body composition, health-related quality of life, depression, and anxiety, as well as their cost-utility.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older.
* Community-dwelling older adults.
* Regular attendance at most sessions (at least 80% attendance).
* Ability to move autonomously, with or without technical assistance.
* Provision of informed consent.

Exclusion Criteria:

* Presence of severe cognitive deficits, assessed by the Pfeiffer test (8 to 10 errors) (Martínez de la Iglesiaa et al., 2001).
* Lack of participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Limited to biological sex.
Enrollment: 240 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
sedentary behavior | From enrollment to the end of the intervention at 12 weeks + 6 months follow-up + 1 year follow-up.
  Change in sedentary behavior mesured by the change in the register pre and post intervention with the activePAL device and the use of sedentary behavior questionaire (SBQ).
  SBQ: Each item rated on a 9-point scale of daily time spent in sedentary activities (0 = none, 8 = ≥6 hours). Total score = sum of minutes across items. Range: 0-3240 minutes/day. Higher scores = worse outcome (more sedentary time). Lower scores = better outcome (less sedentary time).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Blanquerna - Ramon Llull University, Barcelona, Barcelona
  - Universitat Blanquerna, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No